CLINICAL TRIAL: NCT03438370
Title: Outcomes of Differentiated Models of Antiretroviral Treatment (ART) Provision: Multi-Month Dispensing (MMD) of ART in Community ART Distribution for Stable HIV Infected Patients
Brief Title: Outcomes of Differentiated Models of Antiretroviral Treatment (ART) Provision
Acronym: [MMD]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Equip, Lesotho (Other)
Collaborators: Ministry of Health, Lesotho (Other Government); United States Agency for International Development (USAID) (U.S. Federal Agency); Elizabeth Glaser Pediatric AIDS Foundation (Other); Lesotho Network of AIDS Services Organizations (Unknown); National Drugs Service Organisation of Lesotho (Unknown); Chemonics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ID49-2017
Record Dates: First submitted 2017-08-01; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial comparing three different antiretroviral therapy (ART) dispensing strategies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Three monthly ART supply at facilities (No Intervention): Sites at which patients will be provided three monthly ART supply at health facilities.
- Three monthly ART supply at CAGs (Experimental): Sites at which patients will be provided three monthly ART supply at Community ART Groups (CAGs).
  Interventions: Other: Three monthly ART supply at CAGs
- Six monthly ART supply at outreaches (Experimental): Sites at which patients will be provided six monthly ART supply at Community distribution points or outreaches.
  Interventions: Other: Six monthly ART supply at outreaches

INTERVENTIONS:
Other: Three monthly ART supply at CAGs — Sites where three monthly ART supply will be provided at outreaches
  Arms: Three monthly ART supply at CAGs
Other: Six monthly ART supply at outreaches — Sites where six monthly ART will supply will be provided at outreaches
  Arms: Six monthly ART supply at outreaches

SUMMARY:
The aim of this study is to evalulate the effectiveness and cost-effectiveness of three models of ART provision for stable ART patients. The objectives are to measure patient retention, virological suppression, provider and patient costs, cost-effectiveness, and patient acceptability amongst stable patients who receive ART at intervals of three and six months within community distribution models, and to compare these to patients who receive ART directly from the clinic at three month intervals.

Methods

A prospective, parallel, cluster-randomized non-inferiority trial with three study arms will be conducted. 30 Clusters (sites) will be randomized in strata according to geographic location (urban and rural) to the 3 study arms as follows:

* Control arm: sites at which patients will receive three monthly ART supply at the facility (arm 3MF).
* Intervention arm 1: sites at which patients will receive three monthly ART supply in CAGs (arm 3MC)
* Intervention arm 2: sites at which patients will receive six monthly ART supply in the community by a healthcare worker (arm 6MCD).

The study population will consist of stable, HIV-infected adults who have received first-line ART for at least six months, who have a viral load <1000 copies/ml at baseline, and who provide informed consent for inclusion in the study. An average of 192 participants from each study site will be included, with a total sample size of approximately 5760 participants.

The primary outcome is retention in care defined as the proportion of patients remaining in care 12 months after study enrolment, with the hypothesis that patient retention within the intervention arms will be non-inferior compared to the control arm. Retention in care will also be compared between the three arms after 24 months.

The secondary outcomes are:

* Viral suppression: defined as the proportion of patients with virological suppression (<1000 copies/ml) 12 and 24 months after study enrolment;
* Cost of providing ART: defined as the cost per patient of providing ART in each of the three arms (from a provider perspective);
* Cost of retaining a patient: defined as the provider cost per patient retained and provider cost per patient retained with virological suppression in each of the three arms, and the incremental cost-effectiveness ratio for the comparative arms.

DETAILED DESCRIPTION:
Background In 2015, sub-Saharan Africa was still the region most affected by the HIV epidemic, with 25.6 (23.1-28.5) million people living with HIV in 2015. It is estimated that 42% of all people living with HIV (PLHIV) in Lesotho were receiving ART by 2015.The United States Government's President's Emergency Plan for AIDS Relief (PEPFAR) has adopted the goals of 90-90-90 from UNAIDS, and is supporting a swift implementation of the new World Health Organization'sTest and Start guidelines.With these goals, PEPFAR also sets out to reduce new infections by 75% and to attain zero discrimination and stigma for all PLHIV.

To assist countries to reach the goal of universal coverage, EQUIP Innovation for health (a new field support award from the USAID Office of HIV and AIDS that supports innovations in HIV clinical and community-based HIV treatment related services) is evaluating communitybased care, treatment and support models to create an enabling environment for massive scale-up of ART delivery and adherence support. Based on this background, EQUIP and and Elizabeth Glaser Pediatric AIDS Foundation (EGPAF) propose to conduct operational research that seeks to understand and measure the effectiveness of implementing a package of services that include multi-month dispensing (MMD) of ART drugs, Community ART distribution models through Community ART Groups (CAGs) and Community Distribution points and routine viral load monitoring of stable patients in communities of PEPFAR/USAID Lesotho scale-up districts.

The aim of this study is to evalulate the effectiveness and cost-effectiveness of three models of ART provision for stable ART patients. The objectives are to measure patient retention, virological suppression, provider and patient costs, cost-effectiveness, and patient acceptability amongst stable patients who receive ART at intervals of three and six months within community distribution models, and to compare these to patients who receive ART directly from the clinic at three month intervals.

Methods

A prospective, parallel, cluster-randomized non-inferiority trial with three study arms will be conducted. 30 Clusters (sites) will be randomized in strata according to geographic location (urban and rural) to the 3 study arms as follows:

* Control arm: sites at which patients will receive three monthly ART supply at the facility (arm 3MF).
* Intervention arm 1: sites at which patients will receive three monthly ART supply in CAGs (arm 3MC)
* Intervention arm 2: sites at which patients will receive six monthly ART supply in the community by a healthcare worker (arm 6MCD).

Sites for inclusion in the study will be selected at which it is deemed to be feasible to implement multi-month dispensing of ART in the community.

The study population will consist of stable, HIV-infected adults who have received first-line ART for at least six months, who have a viral load <1000 copies/ml at baseline, and who provide informed consent for inclusion in the study. An average of 192 participants from each study site will be included, with a total sample size of approximately 5760 participants. For those sites randomized to the 3MC arm, enrolled participants will be part of a CAG for the duration of the study. For those sites randomized to the 6MCD arm, enrolled participants will be dispensed a 6-month supply of ART in the community by a healthcare worker in between their annual clinical assessments. All participants will have a clinical assessment and viral load testing at the clinic at least annually, and participants will be followed-up for 24 months after enrolment.

The primary outcome is retention in care defined as the proportion of patients remaining in care 12 months after study enrolment, with the hypothesis that patient retention within the intervention arms will be non-inferior compared to the control arm. Retention in care will also be compared between the three arms after 24 months.

The secondary outcomes are:

* Viral suppression: defined as the proportion of patients with virological suppression (<1000 copies/ml) 12 and 24 months after study enrolment;
* Cost of providing ART: defined as the cost per patient of providing ART in each of the three arms (from a provider perspective);
* Cost of retaining a patient: defined as the provider cost per patient retained and provider cost per patient retained with virological suppression in each of the three arms, and the incremental cost-effectiveness ratio for the comparative arms.

Qualitative research will include assessing the acceptability of multi-month dispensing of ART within CAGs and the community from both a patient and healthcare provider perspective. Costs to patients will be compared between the three arms from data derived from patient surveys. In addition, indicators of potential facility level decongestion will be compared between arms, which will include the median facility patient waiting time and average monthly number of patients newly initiated on ART, with data derived from site surveys and routine facility-level data.

This study will follow the ethical considerations specified by the Lesotho National Health Research and Ethics Committee.

The results of the study are expected to inform health policy both nationally and regionally regarding the effectiveness of implementing a package of services consisting of MMD within CAGs and community distribution together with viral load monitoring for stable ART patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and willing and able to provide written informed consent for participation in this study.
* Willing to participate in the multi-month dispensing model that the patient's study site has been randomized to.
* On ART ≥ 6 months with no periods of defaulting from ART since the last viral load result (ART default defined as missing 7 or more consecutive days of ART)
* On first-line ART regimen (substitutions within the first-line regimen prior to the last viral load test are permissible).
* No ARV drug substitutions since the last viral load result < 1,000 copies per ml
* Plasma or dried-blood spot viral load < 1,000 copies/ml in a patient who has been on first-line ART for at least 6 months, with viral load drawn within last 12 months of enrollment while patient is receiving ART

Exclusion Criteria:

* On second-line ART regimen.
* Patients with co-morbidities requiring facility visits more often than 6 monthly.
* ART substitutions since last VL test.
* Diagnosed with a WHO clinical stage 3 or 4 condition within the past 3 months.
* Pregnant or less than 12 months postpartum and breastfeeding mothers.
* Participating in another study that involves dispensing interval, adherence, or retention or involves receiving medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5760 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
retention in care | 12 months
  The proportion of patients remaining in care 12 months after study enrolment

SECONDARY OUTCOMES:
Viral suppression | 12 months
  The proportion of patients with virological suppression (<1000 copies/ml) 12 months after study enrolment
Cost of providing ART | 12 months
  The cost per patient of providing ART in each of the three arms (from a provider perspective)
Cost of retaining a patient | 12 months
  The provider cost per patient retained and provider cost per patient retained with virological suppression in each of the three arms

CONTACTS AND LOCATIONS:
Overall Officials: Iyiola Faturiyele, MBChB, MPH, Principal Investigator — Member, Southern Africa HIV Clinician Society, Johannesburg, South Africa, 2010-present
Locations (1):
- Ha Tlali, Maseru, Lesotho

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WHO. HIV/AIDS: Fact sheet. 2016 [cited 2016 12/12/2016].
- [Background] The Joint United Nations Programme on HIV / AIDS (UNAIDS). Project update. Pac AIDS Alert Bull. 1999;(18):15-6. PMID 12349391
- [Background] Government of Lesotho. National guidelines on the use of antiretroviral therapy for HIV prevention and treatment. In: MOH, editor.2014
- [Background] MOH Lesotho. GLOBAL AIDS RESPONSE PROGRESS REPORT 2015. 2015 Reporting Period: January - December 2014.
- [Background] Guideline on When to Start Antiretroviral Therapy and on Pre-Exposure Prophylaxis for HIV. Geneva: World Health Organization; 2015 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK327115/ PMID 26598776
- [Background] Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV Infection: Recommendations for a Public Health Approach. 2nd edition. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK374294/ PMID 27466667
- [Background] Teck R. Reducing frequency of ARV pick-ups for HIV patients stabilised on ARV treatment 2015.
- [Background] Lesotho Go. Lesotho CAG toolkit In: MOH, editor.2015.
- [Background] Joint United Nations Programme on HIV/AIDS (UNAIDS). COMMUNITY-BASED ANTIRETROVIRAL THERAPY DELIVERY. EXPERIENCES OF MÉDECINS SANS FRONTIÈRES. 2015.
- [Background] World Health Organization. Retention in HIV programmes: defining the challenges and identifying solutions: meeting report, 13-15 September 2011. 2012.
- [Result] Bemelmans M, Baert S, Goemaere E, Wilkinson L, Vandendyck M, van Cutsem G, Silva C, Perry S, Szumilin E, Gerstenhaber R, Kalenga L, Biot M, Ford N. Community-supported models of care for people on HIV treatment in sub-Saharan Africa. Trop Med Int Health. 2014 Aug;19(8):968-77. doi: 10.1111/tmi.12332. Epub 2014 May 28. PMID 24889337
- [Result] Loeliger KB, Niccolai LM, Mtungwa LN, Moll A, Shenoi SV. Antiretroviral therapy initiation and adherence in rural South Africa: community health workers' perspectives on barriers and facilitators. AIDS Care. 2016 Aug;28(8):982-93. doi: 10.1080/09540121.2016.1164292. Epub 2016 Apr 4. PMID 27043077
- [Result] Tiruneh YM, Galarraga O, Genberg B, Wilson IB. Retention in Care among HIV-Infected Adults in Ethiopia, 2005- 2011: A Mixed-Methods Study. PLoS One. 2016 Jun 7;11(6):e0156619. doi: 10.1371/journal.pone.0156619. eCollection 2016. PMID 27272890
- [Result] Rasschaert F, Decroo T, Remartinez D, Telfer B, Lessitala F, Biot M, Candrinho B, Van Damme W. Sustainability of a community-based anti-retroviral care delivery model - a qualitative research study in Tete, Mozambique. J Int AIDS Soc. 2014 Oct 6;17(1):18910. doi: 10.7448/IAS.17.1.18910. eCollection 2014. PMID 25292158
- [Result] Tuller DM, Bangsberg DR, Senkungu J, Ware NC, Emenyonu N, Weiser SD. Transportation costs impede sustained adherence and access to HAART in a clinic population in southwestern Uganda: a qualitative study. AIDS Behav. 2010 Aug;14(4):778-84. doi: 10.1007/s10461-009-9533-2. Epub 2009 Mar 13. PMID 19283464
- [Result] Amanyire G, Wanyenze R, Alamo S, Kwarisiima D, Sunday P, Sebikaari G, Kamya M, Wabwire-Mangen F, Wagner G. Client and provider perspectives of the efficiency and quality of care in the context of rapid scale-up of antiretroviral therapy. AIDS Patient Care STDS. 2010 Nov;24(11):719-27. doi: 10.1089/apc.2010.0108. Epub 2010 Oct 29. PMID 21034243
- [Result] Fay H, Baral SD, Trapence G, Motimedi F, Umar E, Iipinge S, Dausab F, Wirtz A, Beyrer C. Stigma, health care access, and HIV knowledge among men who have sex with men in Malawi, Namibia, and Botswana. AIDS Behav. 2011 Aug;15(6):1088-97. doi: 10.1007/s10461-010-9861-2. PMID 21153432
- [Result] Rollins NC, Becquet R, Orne-Gliemann J, Phiri S, Hayashi C, Baller A, Shaffer N; INSPIRE Team. Defining and analyzing retention-in-care among pregnant and breastfeeding HIV-infected women: unpacking the data to interpret and improve PMTCT outcomes. J Acquir Immune Defic Syndr. 2014 Nov 1;67 Suppl 2:S150-6. doi: 10.1097/QAI.0000000000000355. PMID 25310122
- [Result] Geng EH, Glidden DV, Emenyonu N, Musinguzi N, Bwana MB, Neilands TB, Muyindike W, Yiannoutsos CT, Deeks SG, Bangsberg DR, Martin JN. Tracking a sample of patients lost to follow-up has a major impact on understanding determinants of survival in HIV-infected patients on antiretroviral therapy in Africa. Trop Med Int Health. 2010 Jun;15 Suppl 1(Suppl 1):63-9. doi: 10.1111/j.1365-3156.2010.02507.x. PMID 20586962
- [Result] Roy M, Czaicki N, Holmes C, Chavan S, Tsitsi A, Odeny T, Sikazwe I, Padian N, Geng E. Understanding Sustained Retention in HIV/AIDS Care and Treatment: a Synthetic Review. Curr HIV/AIDS Rep. 2016 Jun;13(3):177-85. doi: 10.1007/s11904-016-0317-9. PMID 27188300
- [Result] Decroo T, Koole O, Remartinez D, dos Santos N, Dezembro S, Jofrisse M, Rasschaert F, Biot M, Laga M. Four-year retention and risk factors for attrition among members of community ART groups in Tete, Mozambique. Trop Med Int Health. 2014 May;19(5):514-21. doi: 10.1111/tmi.12278. Epub 2014 Feb 12. PMID 24898272
- [Result] Marconi VC, Wu B, Hampton J, Ordonez CE, Johnson BA, Singh D, John S, Gordon M, Hare A, Murphy R, Nachega J, Kuritzkes DR, del Rio C, Sunpath H; South Africa Resistance Cohort Study Team Group Authors. Early warning indicators for first-line virologic failure independent of adherence measures in a South African urban clinic. AIDS Patient Care STDS. 2013 Dec;27(12):657-68. doi: 10.1089/apc.2013.0263. PMID 24320011
- [Result] Cohen M, Chen Y, McCauley M, Gamble T, Hosseinipour M, Kumarasamy N, et al., editors. Final results of the HPTN 052 randomized controlled trial: antiretroviral therapy prevents HIV transmission. Journal of the International AIDS Society; 2015: INT AIDS SOCIETY AVENUE DE FRANCE 23, GENEVA, 1202, SWITZERLAND.
- [Result] Ndahimana Jd, Riedel DJ, Mwumvaneza M, Sebuhoro D, Uwimbabazi JC, Kubwimana M, Mugabo J, Mulindabigwi A, Kirk C, Kanters S, Forrest JI, Jagodzinski LL, Peel SA, Ribakare M, Redfield RR, Nsanzimana S. Drug resistance mutations after the first 12 months on antiretroviral therapy and determinants of virological failure in Rwanda. Trop Med Int Health. 2016 Jul;21(7):928-35. doi: 10.1111/tmi.12717. Epub 2016 Jun 13. PMID 27125473
- [Result] Stadeli KM, Richman DD. Rates of emergence of HIV drug resistance in resource-limited settings: a systematic review. Antivir Ther. 2013;18(1):115-23. doi: 10.3851/IMP2437. Epub 2012 Oct 10. PMID 23052978
- [Result] McMahon JH, Elliott JH, Bertagnolio S, Kubiak R, Jordan MR. Viral suppression after 12 months of antiretroviral therapy in low- and middle-income countries: a systematic review. Bull World Health Organ. 2013 May 1;91(5):377-385E. doi: 10.2471/BLT.12.112946. Epub 2013 Feb 21. PMID 23678201
- [Result] Ammassari A, Trotta MP, Shalev N, Marconi P, Antinori A. Beyond virological suppression: the role of adherence in the late HAART era. Antivir Ther. 2012;17(5):785-92. doi: 10.3851/IMP2084. Epub 2012 Mar 13. PMID 22414552
- [Result] Coker M, Etiebet MA, Chang H, Awwal G, Jumare J, Musa BM, Babashani M, Habib AG, Dakum P, Abimiku AG, Charurat ME, Blattner WA, Eng M, Ndembi N. Socio-Demographic and Adherence Factors Associated with Viral Load Suppression in HIV-Infected Adults Initiating Therapy in Northern Nigeria: A Randomized Controlled Trial of a Peer Support Intervention. Curr HIV Res. 2015;13(4):279-85. doi: 10.2174/1570162x13666150407143838. PMID 25845393
- [Result] Fatti G, Shaikh N, Eley B, Grimwood A. Improved virological suppression in children on antiretroviral treatment receiving community-based adherence support: a multicentre cohort study from South Africa. AIDS Care. 2014 Apr;26(4):448-53. doi: 10.1080/09540121.2013.855699. Epub 2013 Nov 11. PMID 24215157
- [Result] Ferrand RA, Briggs D, Ferguson J, Penazzato M, Armstrong A, MacPherson P, Ross DA, Kranzer K. Viral suppression in adolescents on antiretroviral treatment: review of the literature and critical appraisal of methodological challenges. Trop Med Int Health. 2016 Mar;21(3):325-33. doi: 10.1111/tmi.12656. Epub 2016 Jan 10. PMID 26681359
- [Result] Fairall L, Bachmann MO, Lombard C, Timmerman V, Uebel K, Zwarenstein M, Boulle A, Georgeu D, Colvin CJ, Lewin S, Faris G, Cornick R, Draper B, Tshabalala M, Kotze E, van Vuuren C, Steyn D, Chapman R, Bateman E. Task shifting of antiretroviral treatment from doctors to primary-care nurses in South Africa (STRETCH): a pragmatic, parallel, cluster-randomised trial. Lancet. 2012 Sep 8;380(9845):889-98. doi: 10.1016/S0140-6736(12)60730-2. Epub 2012 Aug 15. PMID 22901955
- [Result] Lake S, Kammann E, Klar N, Betensky R. Sample size re-estimation in cluster randomization trials. Stat Med. 2002 May 30;21(10):1337-50. doi: 10.1002/sim.1121. PMID 12185888
- [Result] Xu X, Grossetta Nardini HK, Ruger JP. Micro-costing studies in the health and medical literature: protocol for a systematic review. Syst Rev. 2014 May 21;3:47. doi: 10.1186/2046-4053-3-47. PMID 24887208
- [Result] Scott CA, Iyer H, Bwalya DL, McCoy K, Meyer-Rath G, Moyo C, Bolton-Moore C, Larson B, Rosen S. Retention in care and outpatient costs for children receiving antiretroviral therapy in Zambia: a retrospective cohort analysis. PLoS One. 2013 Jun 28;8(6):e67910. doi: 10.1371/journal.pone.0067910. Print 2013. PMID 23840788
- [Derived] Fatti G, Ngorima-Mabhena N, Tiam A, Tukei BB, Kasu T, Muzenda T, Maile K, Lombard C, Chasela C, Grimwood A. Community-based differentiated service delivery models incorporating multi-month dispensing of antiretroviral treatment for newly stable people living with HIV receiving single annual clinical visits: a pooled analysis of two cluster-randomized trials in southern Africa. J Int AIDS Soc. 2021 Oct;24 Suppl 6(Suppl 6):e25819. doi: 10.1002/jia2.25819. PMID 34713614
- [Derived] Lopes J, Grimwood A, Ngorima-Mabhena N, Tiam A, Tukei BB, Kasu T, Mahachi N, Mothibi E, Tukei V, Chasela C, Lombard C, Fatti G. Out-of-Facility Multimonth Dispensing of Antiretroviral Treatment: A Pooled Analysis Using Individual Patient Data From Cluster-Randomized Trials in Southern Africa. J Acquir Immune Defic Syndr. 2021 Dec 15;88(5):477-486. doi: 10.1097/QAI.0000000000002797. PMID 34506343
- [Derived] Tukei BB, Fatti G, Tiam A, Ngorima-Mabhena N, Tukei VJ, Tshabalala I, Sejana VM, Muzenda T, Mokoroane LM, Sehlabo L, Maotoe T, Mirembe JK, Membe I, Akpan F, Maile K, Faturiyele I, Xulu T, Minior T, Sanne I, Chasela C; for EQUIP Health. Twelve-Month Outcomes of Community-Based Differentiated Models of Multimonth Dispensing of ART Among Stable HIV-Infected Adults in Lesotho: A Cluster-Randomized Noninferiority Trial. J Acquir Immune Defic Syndr. 2020 Nov 1;85(3):280-291. doi: 10.1097/QAI.0000000000002439. PMID 32665460
- [Derived] Faturiyele IO, Appolinare T, Ngorima-Mabhena N, Fatti G, Tshabalala I, Tukei VJ, Pisa PT. Outcomes of community-based differentiated models of multi-month dispensing of antiretroviral medication among stable HIV-infected patients in Lesotho: a cluster randomised non-inferiority trial protocol. BMC Public Health. 2018 Aug 29;18(1):1069. doi: 10.1186/s12889-018-5961-0. PMID 30157896
- See also: UNAIDS. Lesotho: HIV and AIDS estimates. — http://www.unaids.org/en/regionscountries/countries/lesotho